CLINICAL TRIAL: NCT00322270
Title: Phase 3, Multicenter, Multinational, Open-Label Study to Evaluate the Safety and Efficacy of Alfimeprase in Subjects With Occluded Central Venous Access Devices (SONOMA-3)
Brief Title: Safety and Efficacy Study of Alfimeprase in Subjects With Occluded Catheters
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ARCA Biopharma, Inc. (Industry)
Responsible Party: Susan Begelman, MD, Director of Medical Sciences, Nuvelo, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HA008
Record Dates: First submitted 2006-05-03; First posted 2006-05-05 (Estimated); Last update posted 2008-08-15 (Estimated); Status verified 2008-08

CONDITIONS: Thrombosis; Venous Thrombosis; Catheter Occlusion
Keywords: Occluded Central Venous Access Devices; Occluded Catheters; Thrombosis; thrombosis, catheter; alfimeprase; thrombotic occlusion; thrombosis, CVAD; thrombosis, catheters
MeSH Terms: conditions — Thrombosis; Venous Thrombosis | interventions — alfimeprase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Alfimeprase — single-dose of alfimeprase, 10 mg.administered intracatheter to an occluded CVAD

SUMMARY:
To evaluate the safety profile of alfimeprase as assessed by monitoring of adverse events, serious adverse events and major bleeding events for up to 120 minutes following the instillation of study drug to an occluded central venous access device.

DETAILED DESCRIPTION:
Further study details as provided by Nuvelo

ELIGIBILITY:
Inclusion Criteria:

* Must give written informed consent
* Ages 18 or older
* Unable to withdraw at least 3 mL of blood from a central venous access device
* Hemodynamically stable
* Available for follow-up assessments

Exclusion Criteria:

* Inability to infuse at least 2 mL of saline through the catheter
* Catheter placed less than 48 hours prior to detection of occlusion
* Catheter used for hemodialysis or pheresis
* Previous treatment with plasminogen activator for current episode of catheter occlusion
* Less than 18 years of age
* Any evidence of mechanical or nonthrombotic occlusion
* In the opinion of the investigator, subject is at "high risk" for bleeding events of embolic complications, or has a condition for which bleeding constitutes a significant hazard
* Increased risk for drug extravasation
* Pregnant, lactating, or actively menstruating women and women of child-bearing potential who are not using adequate contraceptive precautions (e.g., intrauterine device, oral contraceptives, barrier methods, or other contraception deemed adequate by the investigator)
* Known right-to-left cardiac shunt, patent foramen ovale, or atrial/ventricular septal defect
* Participation in any other study of an investigational device, medication, biologic, or other agent within 30 days before enrollment and until the 30-day follow up visit
* Any other subject feature that in the opinion of the investigator should preclude study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-01

PRIMARY OUTCOMES:
Safety and efficacy | up to120 minutes post study drug dosing

SECONDARY OUTCOMES:
Adverse events, serious adverse events and bleeding events | 24 hours post dosing
Adverse events up to day 30 visit(day 28-45) after instillation of study drug | approximately 28-45 days post dosing

CONTACTS AND LOCATIONS:
Overall Officials: Susan Begelman, M.D., Study Director — ARCA Biopharma, Inc.
Locations (18):
- United States (18):
  - Desert Oasis Cancer Center, Casa Grande, Arizona
  - Cancer Research & Prevention Center, Soquel, California
  - Bethesda Research Center, Boynton Beach, Florida
  - Pasco Hernando Oncology Associates, Brooksville, Florida
  - Mercy Hospital, Miami, Florida
  - Pasco Hernando Oncology Associate, New Port Richey, Florida
  - Medical and Surgical Specialists, Galesburg, Illinois
  - Cancer Center at Blessing Hospital, Quincy, Illinois
  - Kalamazoo Hematology and Oncology, Kalamazoo, Michigan
  - Sparrow Cancer Center, Lansing, Michigan
  - Comprehensive Cancer Care Clinic, Jefferson City, Missouri
  - The Center for Cancer Care and Research, St Louis, Missouri
  - UMDNJ-Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Dakota Cancer Institute, Fargo, North Dakota
  - Gabrail Cancer Center, Canton, Ohio
  - Hematology/Oncology Consultants, Inc., Columbus, Ohio
  - Texas Oncology, P.A., Dallas, Texas
  - Carilion Gynecology/Oncology, Roanoke, Virginia